CLINICAL TRIAL: NCT05575934
Title: Management of Transitory Loss of Consciousness and Syncopes in the Emergency Department
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: EI22MG0908
Record Dates: First submitted 2022-10-04; First posted 2022-10-12 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Syncope; Unconscious State
Keywords: transient loss of consciousness; syncope; emergency department
MeSH Terms: conditions — Syncope; Unconsciousness; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to examine the clinical presentations, the diagnostic tests performed and the management of patients presenting with transient loss of consciousness (TLOC)

The main questions it aims to answer are:

* prevalence of TLOC
* prevalence of different diagnoses leading to TLOC Demographic, clinical, paraclinical and biological data will be collected from the emergency medical file

DETAILED DESCRIPTION:
Patients over the age of 18 presenting to the University Hospital of Clermont-Ferrand emergency department for transient loss of consciousness of syncopal or undifferentiated origin will be include. Their non-opposition will be sought.

Demographic, clinical, paraclinical and biological data will be collected from the emergency medical file.

No visit is planned after the passage to the emergency room.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 presenting to the Clermont-Ferrand University Hospital emergency department for transient loss of consciousness of syncopal or undifferentiated origin

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients presenting to the emergency room of the CHU de Clermont-Ferrand with a transient loss of consciousness of syncopal or undifferentiated origin will be included once the non-objection has been collected.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-10-03 (Actual); Primary Completion 2023-03-25 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
prevalence of transient loss of consciousness in emergency department | through the study duration, an average of 6 months
  Percentage of TLOC in emergency department
prevalence of different diagnoses leading to transient loss of consciousness | through the study duration, an average of 6 months
  Percentage of different diagnoses leading to transient loss of consciousness

SECONDARY OUTCOMES:
prevalence of different clinical presentations of loss of consciousness | through the study duration, an average of 6 months
  Percentage of different clinical presentations of loss of consciousness
Prevalence of the various diagnostic tests carried out and the treatment of patients presenting for transient loss of consciousness | through the study duration, an average of 6 months
  Percentage of the various diagnostic tests carried out and the treatment of patients presenting for transient loss of consciousness

CONTACTS AND LOCATIONS:
Overall Officials: Fares Moustafa, MD, PhD, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France